CLINICAL TRIAL: NCT00737347
Title: Prevention of Weight Gain in Adult Patients With Type 2 Diabetes Treated With Pioglitazone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Robert F. Kushner, MD, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0309-015
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: type 2 diabetes; obesity; weight gain; thiazolidinediones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): usual care. Subjects had one 90 minute visit with registered dietitian
- 2. (Active Comparator): Standard care. Subjects had 4 sessions with registered dietitian
  Interventions: Behavioral: Lifestyle modification
- 3 (Active Comparator): Intensive care. subjects had 10 visits with registered dietitian
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Behavioral: Lifestyle modification — lifestyle intervention includes meal planning, food preparation, food label reading, dining out, and physical activity counseling
  Other Names: lifestyle behavioral counseling
  Arms: 2.; 3

SUMMARY:
The purpose of the study is to investigate the effectiveness of three lifestyle treatment programs varying in level of intensiveness on prevention of pioglitazone-induced weight gain and to measure the composition of the change in body weight.

DETAILED DESCRIPTION:
The three lifestyle interventions were usual care (1 visit), standard care (4 total visits) and intensive care (10 total visits)

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with BMI 27 or greater, glycated hemoglobin 7% or greater

Exclusion Criteria:

* insulin treated

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-09; Primary Completion 2007-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
change in body weight | 24 weeks

SECONDARY OUTCOMES:
change in body composition | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Kushner, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital Wellness Institute, Chicago, Illinois, United States